CLINICAL TRIAL: NCT01562457
Title: A Randomised, Open-label, Multi-centre Trial Investigating the Intra-subject Variability of ROTEM® and TEG® Parameters Following Two Intravenous Administrations of the Same Dose of Activated Recombinant Factor VII (rFVIIa/NovoSeven®) in Haemophilia Patients in a Non-bleeding State
Brief Title: Intra-subject Variability Following Administrations of Activated Recombinant Human Factor VII in Haemophilia Patients in a Non-bleeding State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1731-1668; 2005-000891-42 (EudraCT Number)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Medium dose (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- High dose (Experimental)
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — Administered as a single dose. Injected as a slow intravenous injection over 2 minutes (from start to completion of injection)

SUMMARY:
This trial is conducted in Asia and Europe. The aim of this trial is to evaluate the intra-subject variability of thromboelastographic parameters (TEG® and ROTEM®) following two administrations of activated recombinant human factor VII in haemophilia patients in a non bleeding state.

The TEG® parameters are: R time (Reaction Time), K time (K Time (arbitrary measurement)), a (a angle), MA (Maximum Amplitude) and LY30 (Lysis 30 min after MA) while the ROTEM® parameters are: CT (Clotting Time), CFT (Clot Formation Time), a (a angle), MCF (Maximum Clot Firmness) and LI60 (Lysis index 60 min after CT).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of congenital haemophilia A or B with a FVIII:C (Activated Coagulation Factor VIIa Clotting activity) or FIX:C (Coagulation Factor IX Clotting activity) one stage activity, respectively, at less than 5% of normal (based on medical records) plus/minus inhibitors (a positive inhibitor status defined as 0.6 Bethesda units)
* Non-bleeding state (i.e. no clinical manifestation of active bleed) at the time of administration of trial product

Exclusion Criteria:

* Known or suspected allergy to trial product or any of its components or to related products
* Known clinically relevant coagulation disorders or insufficiencies other than congenital haemophilia A or B
* Platelet count below 50,000 platelets/mcL
* Received any haemostatic treatment (e.g. Feiba) within the last 7 days prior to administration of trial product, except for activated recombinant human factor VII

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-11; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
TEG® (Thromboelastography) parameters after dosing of trial product
ROTEM® (Thromboelastometry) parameters after dosing of trial product

SECONDARY OUTCOMES:
TEG® parameters obtained from blood samples spiked ex vivo with activated recombinant human factor VII
ROTEM® parameters obtained from blood samples spiked ex vivo with activated recombinant human factor VII
Serious adverse events and non-serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Lille, France
- München, Germany
- Tel Litwinsky, Israel

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com